CLINICAL TRIAL: NCT04456231
Title: Effect of the Additional Use of a QR Code for More Effective Patient Education and High-quality Bowel Preparation in the Outpatient Setting
Brief Title: QR Code for Endoscopic Bowel Preparation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Prof. Helmut Neumann, University Professor Dr. med., Johannes Gutenberg University Mainz
Other Study IDs: 126
Record Dates: First submitted 2020-06-16; First posted 2020-07-02 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Quality Standards in Colonoscopy; Patient Education; Acceptance of Bowel-preparation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- QR Code: Patients will drink 1 Liter of Plenvu and 1 Liter of water or tea in preparation for endoscopy according to endoscopy Guidelines. In Addition, this Group will receive a health app for better preparation and more Information regarding preparation and endoscopy itself.
  Interventions: Drug: Plenvu
- no QR Code: Patients will drink 1 Liter of Plenvu and 1 Liter of water or tea in preparation for endoscopy according to endoscopy Guidelines. This Group will have no app and will have to receive Information in traditional ways.
  Interventions: Drug: Plenvu

INTERVENTIONS:
Drug: Plenvu — Patients will receive Plenvu for preparation of endoscopy

SUMMARY:
Patients presenting for colonoscopy at one of the participating centers will be asked to participate in the present study after careful evaluation of inclusion and exclusion criteria. Before inclusion, all patients have to sign the written informed consent. All participating patients will receive PLENVU, a well-known and approved bowel preparation agent. Patients are randomly assigned in two groups. Patients in group 1 are informed in traditional way on how to use the bowel preparation agent. This way includes discussion with the physician and nurse on how to use the bowel preparation agent and a written documentation, highlighting the individual steps again. Patients in group 2 will receive in addition a QR-code referring to an App, available for free in all App stores, explaining to the patient in detail when and how to use the bowel preparation agent. The patient is receiving the same questionnaire (please see attached) in both groups and asked to bring the filled form on the day of the examination. Endoscopy is performed in standard way and effectiveness of the bowel preparation is specifically highlighted by the physician on the documentation report. Finally, data is analyzed regarding effectiveness of the QR code regarding patient satisfaction, acceptability and quality of the bowel preparation.

DETAILED DESCRIPTION:
Patient education is of paramount importance for high acceptance and an adequate bowel preparation. Using the QR code directly referring to the App for bowel preparation with PLENVU might accelerate the discussion between the medical doctor and the patient and might also improve the acceptance rate of the patients for the bowel preparation finally leading to a more enhanced and effective bowel-preparation.

Patients undergoing screening or surveillance endoscopy will be prospectively included and randomly assigned to one of the following groups: Group 1: App; Group 2: no-App Study end points addressed below are prospectively assessed and evaluated for any significant changes.

ELIGIBILITY:
Inclusion Criteria:

* • Screening or surveillance colonoscopy

  * Age 18-85 years
  * Written informed consent

Exclusion Criteria:

* • Pregnancy or lactating

  * Lower gastrointestinal bleeding with hemodynamic instability
  * Bowel obstruction
  * ASA >3
  * Not sufficiently corrected anticoagulation disorders
  * Plenvu must not be taken:

    * if you are allergic (hypersensitive) to the active ingredients or any of the other ingredients of this medicine;
    * if you have a blockage (obstruction) in the digestive tract.
    * if you have a breakthrough (perforation) in the wall of the digestive tract;
    * if you suffer from intestinal obstruction (Ileus);
    * if you suffer from a disturbance of gastric emptying (e.g. gastroparesis, gastric retention);
    * if you suffer from phenylketonuria. Phenylketonuria is a congenital metabolic disease in which phenylalanine cannot be processed by your body. Plenvu contains aspartame as a source of phenylalanine;
    * if you suffer from glucose-6-phosphate dehydrogenase deficiency;
    * if you suffer from acute colon enlargement (toxic megacolon).
  * Warnings and precautions

    o You should tell your doctor about the following circumstances before taking Plenvu:
  * if you have heart problems and/or arrhythmias;
  * if you have kidney problems and/or suffer from dehydration;
  * if you have stomach or intestinal problems, including intestinal inflammation;
  * if you have difficulty or discomfort when swallowing liquids;
  * if you have high or low levels of electrolyte (e.g. sodium, potassium);
  * if you have other diseases (e.g. convulsions).
  * Pregnancy and lactation o There are no data on the use of Plenvu during pregnancy or lactation and is therefore not recommended.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: patients receiving traditional information how to prepare the colon Group 2: patients receiving in addition a QR-code referring to an App, available for free in all App stores, explaining to the patient in detail when and how to use the bowel preparation agent
Sampling Method: Probability Sample
Enrollment: 404 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Standard (BBPS) | 1 day
  Bowel preparation according to international Standard, 1 is bad, 9 is very good, how many patients can Achieve BBPS with 9?
Adenoma detection rate (ADR) | 1 day
  How many adenomas will be detected during endoscopy
Polyp detection rate (PDR) | 1 day
  How many polyps will be detected during endoscopy
time exposure to explain bowel preparation | 1 day
  How much time will patients Need for preparation and how much time for discussing with the doctors

SECONDARY OUTCOMES:
Number of patients who are satisfied with preparation | up to 1 month
  How will doctors and patients like preparation with Plenvu and QR Code
Number of patients who Accept to repeat the examination (surveillance) | up to 1 month
  How many patients will come back for another endoscopy
cecal intubation rate | 1 day
  How many endoscopies will reach the ceacum
procedure time | 3 hours
  How Long will endoscopy take compared to Standard technique

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, Prof. Dr., Principal Investigator — University Medical Center Mainz
Locations (1):
- Dr. Helmut Neumann, Bad Salzuflen, Northrine-Westfalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Preliminary results for DDW (Deadline Dec, 1st, 2020) .
  Publication date:
  * Preliminary data 2020 for: DDW 2021 (Deadline Dec. 1st), preliminary data will be available for Norgine for DGVS (Germany) and APDW (Malaysia).
  * Final data: Submission 2021 for DDW, ESGE Days, UEGW, DGVS, APDW
  * Final manuscript: Gut -> Am J Gastro -> Endoscopy
Supporting Information: Study Protocol, ICF
Time Frame: First Data: January 2021 full Data: December 2021
Access Criteria: Abstracts and Publication